CLINICAL TRIAL: NCT03865355
Title: Unique Blood and CSF Metabolic Profile Association With Gliomas in Adults
Brief Title: Blood and Cerebrospinal Fluid Metabolomic Profile in Glioma Patients
Status: Completed | Type: Observational
Sponsor: Novosibirsk State University (Other)
Collaborators: FSBI "Federal Neurosurgical Center" Novosibirsk, Russia (Unknown); Novosibirsk Research Institute of Traumatology and Orthopaedics n.a. Ya.L. Tsivyan (Other Government)
Responsible Party: Sponsor
Other Study IDs: MetGlio/19
Record Dates: First submitted 2019-02-26; First posted 2019-03-06 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Glioma; Glioblastoma Multiforme
Keywords: Metabolomic profile; Biomarkers
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, cerebrospinal fluid (CSF)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1 / High grade Glioma: Cohort 1:
  1. Histologically confirmed high-grade glioma (grade III and grade IV (glioblastoma (GBM)))
  2. Planned treatment (surgery followed by radiation therapy (RT) alone or Chemotherapy alone or a combination of RT/Chemotherapy)
  Interventions: Other: Non- interventional
- Cohort 2 / Low grade Glioma: Cohort 2:
  1. Histologically confirmed low-grade (grade I/II) glioma
  2. Planned treatment either expectant monitoring or surgery followed by RT alone or Chemotherapy alone or a combination of RT/Chemotherapy
  Interventions: Other: Non- interventional
- Cohort 3 / Conditionally healthy volunteers: Cohort 3:
  1. No oncological disease was diagnosed
  2. Planned treatment (reconstructive surgery after craniofacial trauma)
  Interventions: Other: Non- interventional

INTERVENTIONS:
Other: Non- interventional — Translational, observational study

SUMMARY:
This is an exploratory, non-interventional and translational clinical study. The aim of this study is to analyze blood and cerebrospinal fluid metabolomic profile in glioma patients.

DETAILED DESCRIPTION:
The analysis of metabolic profile in the plasma and CSF could become the new less invasive approach in the establishing diagnosis as well as an important prognostic factor in patients with glioma. The researches will assess the blood and CSF metabolic profile in patients with different types of gliomas as well as in patient without ones. This can help to find new biomarkers for low- and high-grade gliomas correlating with patient outcomes.

Blood and CSF samples will be collected from patients with suspected newly diagnosed low-grade (I-II) or high-grade (III-IV) gliomas as well as from patients who have hospitalized for reconstructive surgery after craniofacial trauma. All samples will be collected before any surgical intervention and at various follow-up time points until progression or death. The results of the study are planned to be translated into the hospital setting as support to other diagnostics procedures and to the differential diagnosis between glioma grades.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with suspected newly diagnosed glioma (grade I, II, III or glioblastoma) with planned surgical intervention (resection or biopsy).
2. Patient aged 18 years or older
3. Patients have to be able to give informed consent

Exclusion Criteria:

1. Prior Radiotherapy to the central nervous system
2. Prior Chemotherapy within the last 5 years
3. Any prior central nervous system malignancy
4. Any surgery during last 6 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with suspected newly diagnosed glioma with planned surgical intervention will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Metabolic phenotype of glioma patients | 5 years
  Plasma and CSF aminoacids, acylcarnitines, and other metabolites in glioma patients compared to conditionally healthy volunteers by high-performance liquid chromatography coupled with tandem mass spectrometry.

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  Time between date of diagnosis and date of death
Progression free survival (PFS) | 5 years
  Time between date of diagnosis and date of disease progression

CONTACTS AND LOCATIONS:
Locations (1):
- Novosibirsk State University, Novosibirsk, Novosibirsk Oblast, Russia